CLINICAL TRIAL: NCT02616237
Title: Effects of a Facebook-based Weight Loss Programme for Obese Adults in Hong Kong
Brief Title: A Facebook-based Weight Loss Programme for Obese Adults in Hong Kong
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, LAI Kam Wa, Senior Manager, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20131213002
Record Dates: First submitted 2015-11-24; First posted 2015-11-26 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Obesity
Keywords: Chinese population; acupressure; physical activity; nutrition; Facebook
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): Lifestyle Intervention: The interventions include participation in a private research group on Facebook for health education, self monitoring and social support. Participants will receive 12 weekly lessons related to nutrition, physical activity, Chinese food therapy, acupressure, weight loss. A registered nutritionist and a registered Chinese medicine practitioner will join the Facebook group as health partners. Both of them are also registered nurses.
  Besides the Facebook contents, the participants will also receive government printed health information on healthy eating, physical activity, obesity and cancers.
  Interventions: Behavioral: Lifestyle Intervention
- Control Group (No Intervention): The participants randomized into the Control Group will only receive government printed health information on healthy eating, physical activity, obesity and cancers.

INTERVENTIONS:
Behavioral: Lifestyle Intervention — East-meets-West Lifestyle Intervention elements include nutrition and exercise from the Western perspective, food therapy and acupressure from the Traditional Chinese Medicine perspective, self-monitoring, and motivational videos of successful stories from working colleagues. The group participants in the Facebook are encouraged to post their health behaviors and questions, self-monitor, pledge for weight loss, seek social support and interact with health partners and other participants.
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to determine the feasibility and efficacy of a 6-month weight loss intervention program for obese working adults through a popular social networking site - Facebook.

DETAILED DESCRIPTION:
Obese individuals often are at higher risk for developing non-communicable diseases such as diabetes and cardiovascular disease. The regular physical activity, healthy diet and social support have been shown to be beneficial for weight loss.

This is a two-arm parallel design randomized controlled trial for 6 months. Participants who completed the baseline assessment will be randomly allocated, after stratified by gender, to either a control group or Facebook-based intervention group. The control group will receive information on healthy eating, physical activity, obesity and cancer via three government printed health pamphlets. In addition to the government health pamphlets, the intervention group will receive a programme delivered through Facebook.

The interventions include participation in a private research group on Facebook for health education, self monitoring and social support. Participants will receive 12 weekly lessons related to nutrition, physical activity, Chinese food therapy, acupressure, weight loss. A registered nutritionist and a registered Chinese medicine practitioner will join the Facebook group as health partners. Both of them are also registered nurses.

Data collection will be carried out at baseline, 3 months and 6 months. Each time, both groups will complete online questionnaires and attend in-person anthropometric measurements

ELIGIBILITY:
Inclusion Criteria:

* university full-time employees;
* age 18 to 60 years,
* BMI of 25 to 40 kg/m2,
* have access to Internet and Facebook;
* able to communicate in both English and Chinese at F.5 secondary school level or above.
* agree to communicate with Internet, email, Facebook group and respect privacy.

Exclusion Criteria:

* Smoker;
* an unstable medical or mental status;
* history of myocardial infarction or stroke, or cancer in the past 5 years;
* orthopedic or joint problems that would prohibit exercise;
* in treatment for alcohol or drug dependency;
* an eating disorder;
* pregnant, breastfeeding, or planning on becoming pregnant within the next 6 months;
* use of medication that might affect body weight;
* a recent weight loss of more than 4.5 kg in the previous 6 months;
* currently participating in a weight loss program;
* organic obesity;
* unable to attend assessments or increase physical activity.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2014-04; Primary Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Changes in body weight | Measures are done in three time points: baseline, 3 months and 6 months
  Weights will be taken in light clothes without shoes using a digital scale
Changes in Body Mass Index | Measures are done in three time points: baseline, 3 months and 6 months
  Height will be taken at baseline using a wall-mounted stadiometer. BMI will be calculated as weight (kg)/height (m2)
Changes in waist circumference | Measures are done in three time points: baseline, 3 months and 6 months
  Waist circumference will be measured by using an inelastic tape measure

SECONDARY OUTCOMES:
Changes in Stages of Change | Measures are done in three time points: baseline, 3 months and 6 months
  A 5-item questionnaire will be used to categorize participants into stages of change (pre-contemplation, contemplation, preparation, action, maintenance)
Changes in weight self-efficacy | Measures are done in three time points: baseline, 3 months and 6 months
  Self-efficacy for weight loss will be assessed by using a 20-item Weight Efficacy Lifestyle Questionnaire (WEL).
Changes in physical activity self-efficacy | Measures are done in three time points: baseline, 3 months and 6 months
  A questionnaire of perceived confidence to engage in physical activity under a variety of circumstances on a 5-point Likert scale will be used.
Changes in weight decisional balance | Measures are done in three time points: baseline, 3 months and 6 months
  A 20-item questionnaire of perceived pros and cons of weight loss on a 5-point Likert scale. The balance of the two scores >0 indicate more advantages than disadvantages to weight loss
Changes in social support | Measures are done in three time points: baseline, 3 months and 6 months
  A questionnaire will be used to measure the perceived support and sabotage from friends and family for healthy eating and physical activity
Changes in dietary intake of fruits and vegetables | Measures are done in three time points: baseline, 3 months and 6 months
  A questionnaire will be used to assess self-reported intake of fruits and vegetables in terms of portion size and frequency
Changes in physical activity | Measures are done in three time points: baseline, 3 months and 6 months
  The International Physical Activity Questionnaire will be used to assess the changes in physical activity

CONTACTS AND LOCATIONS:
Overall Officials: WanChaw SHAE, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No